CLINICAL TRIAL: NCT03357705
Title: Effectiveness of Different Alveolar Preservation Procedures in the Upper Molar Zone in Limiting the Need to Elevate the Maxillary Sinus to Allow the Placement of Dental Implants: a Prospective Cohort Multicentre Clinical Study.
Brief Title: Effectiveness in Limiting the Need to Elevate the Maxillary Sinus
Acronym: SO-GHI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Piezosurgery Academy (Other)
Responsible Party: Principal Investigator, Mr. Claudio Stacchi, DDS, MSc, President of the International Piezosurgery Academy, International Piezosurgery Academy
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SO-GHI
Record Dates: First submitted 2017-11-24; First posted 2017-11-30 (Actual); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Alveolar Bone Loss
Keywords: alveolar ridge preservation
MeSH Terms: conditions — Alveolar Bone Loss | interventions — Septodont

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- synthetic (Experimental): alveolar ridge preservation with synthetic bone
  Interventions: Procedure: alveolar ridge preservation with synthetic bone
- collagen (Active Comparator): alveolar ridge preservation with bovine collagen
  Interventions: Procedure: alveolar ridge preservation with bovine collagen

INTERVENTIONS:
Procedure: alveolar ridge preservation with synthetic bone — after tooth extraction
  Other Names: Ghimas
  Arms: synthetic
Procedure: alveolar ridge preservation with bovine collagen — after tooth extraction
  Other Names: Septodont
  Arms: collagen

SUMMARY:
The aim of the present study is to evaluate the effectiveness of different alveolar preservation procedures performed at the time of extraction of the first or second upper molar in avoiding a maxillary sinus elevation or at least limiting the size, to allow the insertion of dental implants. The residual bone height will be radiographically evaluated on the sinus sinus floor at the time of extraction and after 6 months by comparing the cases where alveolar preservation is performed using a nanocrystalline synthetic hydroxyapatite graft (group A) with cases where the procedure of alveolar preservation is performed using bovine collagen sponge (group B).

DETAILED DESCRIPTION:
Bone resorption and contraction of bone volumes are physiologically occurring after the extraction of any dental element. This reabsorption of the alveolar process results in a reduction in the size of the alveolar crest both in width and in height. Numerous studies have attempted to quantify the size and timing of contraction of bone volumes after a dental flotation. The data reported in the literature show an average horizontal reduction of about 2.5 mm, which appears more marked by the vestibular side than the palatal one. The vertical contraction of the crest is estimated at 25-30%, with bone loss of 1-2 mm and a soft contraction of soft tissues of about 2 mm. In the area of the first and second upper molars, however, the total contraction of the alveoli is greater because the residual crest at the insertion of the implant would have undergone a double reduction, namely from the coronal side with the mechanisms just indicated, but also from the apex , for maxillary sinus pneumonia due to the absence of dental element6. For this reason, insertion of an implant in this area may be difficult due to an inadequate height of the remaining bone, which necessitates a bone regeneration procedure, ie a maxillary sinus elevation. This procedure allows you to regain the abdominal apex lost and the insertion of adequate lengths. In the presence of satisfactory residual bone height, maxillary sinus breast can be performed crestally, while in more markedly atrophic cases, especially in the presence of anatomically wide breasts, a side-by-side approach is preferable.

Various grafting materials have been used to perform alveolar retention with the aim of limiting the contraction of bone volumes and improving bone formation: autologous bone, homologous bone and bone substitutes of heterologous origin or alloplastic.

The use of autologous bone in alveolar preservation was soon abandoned for bone marrow morbidity, especially when deciding to use a donor site other than the extraction area. The homologous bone, although showing excellent results, is still to date problematic use in Italy. The heterologous grafts have been widely used for alveolar preservation; however, especially if bovine bone is used, significant percentages of graft (up to 25%) are histologically observable at 9 months from graft.

For these reasons, in this study it was decided to use as a graft in Group A a synthetic material (nanocrystalline synthetic hydroxyapatite) and in group B a collagen of bovine origin.

Bovine collagen, while having reduced dimensional stability over time, has the advantage of contributing to stabilizing the clot, an essential basis for bone healing, and is completely replaced by newly formed tissue in a short time. Synthetic hydroxyapatite, used as a biomaterial, has shown ability to stimulate osteoconduction and is slowly but completely replaced over time by newly formed bone, thus providing a great capacity for maintaining volumes.

Moreover, nanostructured porous hydroxyapatite appear to favor adhesion of bone matrix proteins and promote differentiation of osteogenetic cells. Although the nanocrystalline hydroxyapatite in a silica gel matrix has already been successfully tested as a clotting material in the maxillary sinus, the behavior of pure sintered nano-hydroxyapatite granules has not yet been evaluated in terms of osteoconductive potential and dimensional stability in time at post-mining sites.

ELIGIBILITY:
Inclusion Criteria:

1. indication for extraction of the first or second upper molar, based on a thorough diagnosis and treatment plan;
2. "three-rooted" anatomy of the first or second upper molar to be extracted so that it can have an inter-radicular septum that allows a precise measurement of the height of the bone ridge from the septum itself and from the walls of the 3 alveoli to the floor of the maxillary sinus;
3. Extraction of intercalate molar or last arch element;

Exclusion Criteria:

1. Anatomy of the molar with unique root or fused roots
2. contextual extraction of the molar and one or more contiguous elements
3. apical lesions with a diameter of> 3 mm or cystic lesions with respect to the element to be extracted
4. root fracture which has produced resorption or bone fenestration

1) acute myocardial infarction in the last six months; 2) uncontrolled clotting disorders; 3) uncontrolled diabetes (HBA1c> 7.5%); 4) radiotherapy in the head / neck district for the last 24 months; 5) immunocompromise (eg HIV infection or chemotherapy over the last 3 years); 6) treatment in progress or with bisphosphonates via e.v .; 7) autoimmune diseases in chronic therapy with methotrexate or other immunosuppressive drugs; 8) allergy to bovine collagen; 9) psychological or psychiatric problems; 10) abuse of alcohol or drug use; 11) uncontrolled periodontal disease;

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-10-31 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-12-28 (Actual)

PRIMARY OUTCOMES:
radiographic distance between crestal bone and implant platform | 6 months after surgery
  necessity of sinus floor regeneration

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Stacchi, Dr, Study Director — Piezosurgery Academy
Locations (1):
- Piezosurgery Academy, Parma, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carlsson GE, Bergman B, Hedegard B. Changes in contour of the maxillary alveolar process under immediate dentures. A longitudinal clinical and x-ray cephalometric study covering 5 years. Acta Odontol Scand. 1967 Jun;25(1):45-75. doi: 10.3109/00016356709072522. No abstract available. PMID 5233859
- [Background] Sharan A, Madjar D. Maxillary sinus pneumatization following extractions: a radiographic study. Int J Oral Maxillofac Implants. 2008 Jan-Feb;23(1):48-56. PMID 18416412